CLINICAL TRIAL: NCT04326946
Title: International Alfapump Cohort Study: in Patients With Refractory Ascites Due to Liver Cirrhosis or Malignant Ascites With a Life Expectancy of 6 Months or Less
Brief Title: International Alfapump Cohort Study
Acronym: TOPMOST
Status: Active, not recruiting | Type: Observational
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-AAR-012
Record Dates: First submitted 2018-06-25; First posted 2020-03-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Liver Cirrhoses; Malignant Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Biobanking of urine, ascites and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Alfapump — alfapump implementation

SUMMARY:
This Registry is designed to follow patients who have been implanted with an alfapump system, which is a newly marketed product from Sequana Medical AG, a Swiss Medical Device company.

DETAILED DESCRIPTION:
In a real-world setting, all patients implanted with an alfapump system according to it's intended use, not participating in another clinical study in which the alfapump is studied.

ELIGIBILITY:
Inclusion Criteria:

* All patients implanted with an alfapump are eligible for this registry

Exclusion Criteria:

* Patients younger than 18 years
* Pregnancy
* Inability to operate the Smart Charger to recharge the alfapump
* Participating in another study in which the alfapump is studied

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The TOPMOST will target to include, in a real-world setting, all patients implanted with an alfapump system as per intended use, not participating in another clinical study in which the alfapump is being evaluated.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient survival at 6 months post implant | 6 months post-implant
  The primary outcome will be patient survival with a functional alfapump system at 6 months.

SECONDARY OUTCOMES:
To assess occurrence of (major) reportable events. | 2 years
  Reportable events are defined as any events per the definition in 9.1 and classified as renal event, variceal bleeding, hepatic encephalopathy an infection or assessed as related (not classified "improbable related" or "cannot be attributed" per the definitions below) to; the implant procedure, device or therapy by the treating physician.
To assess safety at 1-month post implant for procedure related incidents. | 1 month post implant
  o Occurrence of adverse events considered related to implant, product or therapy by the treating physician
Clinical impact on liver and renal function in liver & renal blood lab panel | 2 years
  Clinical impact as assessed by changes in Prealbumin
Clinical impact on liver and renal function in liver & renal blood lab panel | 2 years
  Clinical impact as assessed by changes in Albumin.
Clinical impact on liver and renal function in liver & renal blood lab panel | 2 years
  Clinical impact as assessed by changes in eGFR.
Clinical impact on liver and renal function in liver & renal blood lab panel | 2 years
  Clinical impact as assessed by changes in createnine.
Impact of the alfapump on ascites symptoms related quality of life | 2 years
  Ascites Questionnaire (pre implant & at each visit after the first month post implant)
Impact of the alfapump on ascites symptoms related quality of life | 2 years
  SF-36 (pre implant at each visit after the first month post implant)
Impact of the alfapump on ascites symptoms related quality of life on patient activity | 1 week pre-implant, Day 0 Implant, 4 weeks-, 8 weeks-, 16 weeks-, 24 weeks- and 48 weeks post implant
  Assess change in physical activity pre- and post implant To assess daily activity and stress level of patients for up to 48 weeks following implant
Impact of the alfapump on ascites symptoms related quality of life on patient activity | 1 week pre-implant, Day 0 Implant, 4 weeks-, 8 weeks-, 16 weeks-, 24 weeks- and 48 weeks post implant
  Assess change in physical activity pre- and post implant To assess and evaluate sleep of patients for up to 48 weeks following implant
Impact of the alfapump on ascites symptoms related quality of life on patient activity | 1 week pre-implant, Day 0 Implant, 4 weeks-, 8 weeks-, 16 weeks-, 24 weeks- and 48 weeks post implant
  Assess change in physical activity pre- and post implant
  1. To assess daily activity and stress level of patients for up to 48 weeks following implant
  2. To assess and evaluate sleep of patients for up to 48 weeks following implant
  3. To assess patient's abdominal pain/discomfort, appetite, satiety, and tiredness
  4. To assess objective stress and inflammation parameters
Impact of the alfapump on ascites symptoms related quality of life on patient activity | 1 week pre-implant, Day 0 Implant, 4 weeks-, 8 weeks-, 16 weeks-, 24 weeks- and 48 weeks post implant
  Assess change in physical activity pre- and post implant To assess patient's abdominal pain/discomfort, appetite, satiety, and tiredness
Impact of the alfapump on ascites symptoms related quality of life on patient activity | 1 week pre-implant, Day 0 Implant, 4 weeks-, 8 weeks-, 16 weeks-, 24 weeks- and 48 weeks post implant
  Assess change in physical activity pre- and post implant To assess objective stress and inflammation parameters
Clinical impact on ECOG | 2 years
  change in ECOG performance scale pre- and post implant

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Gottardi, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Universitätsklinikum Leipzig, Leipzig, Germany
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
To be decided